CLINICAL TRIAL: NCT06118892
Title: Post-Market Evaluation of the MISHA® Knee System for Symptom Relief in Subjects With Medial Knee Osteoarthritis
Brief Title: MISHA Post-Market Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP0009
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MISHA Knee System (Experimental)
  Interventions: Device: MISHA Knee System

INTERVENTIONS:
Device: MISHA Knee System — The MISHA Knee System is an extra-capsular knee implant intended to reduce loads on the medial knee. The implant consists of an absorber located between bases fixed with locking screws to the medial cortices of the distal femur and proximal tibia. The implant shares the load with the medial knee joint and articulating ball-and-sockets allow the device to accommodate the natural motions of the knee.
  Other Names: Implantable Shock Absorber (ISA)

SUMMARY:
Prospective evaluation of the safety and effectiveness of the MISHA Knee System.

The study will collect data on the procedural and long-term adverse events, WOMAC pain and function scores, KSS satisfaction, subsequent surgical interventions, BMI levels, range of motion, UCLA activity level of the subjects, and perform radiographic/x-ray evaluations at clinical visits through 5 years post-procedure.

The primary analysis of this study is freedom from device- and procedure-related SSIs at five (5) years post-implantation.

This study will also assess device performance in subjects with intact and retained devices and subjects with devices removed prior to study termination and freedom from conversion to arthroplasty through 5 years.

Study subjects will be followed over a five-year post-implant period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects aged 25 to 65 years at time of index procedure
2. Body Mass Index (BMI) of < 35
3. Activity exacerbated knee pain isolated to the medial compartment and not global in nature
4. WOMAC pain ≥ 40
5. Failed non-operative OA treatment

Key Exclusion Criteria:

1. Large medial osteophyte(s) or considerable extruded meniscus that may interfere with the placement or function of the device
2. Poor bone quality (e.g., bony erosion, osteopenia, osteoporosis)
3. Ligamentous instability
4. Active or recent knee infection
5. Inflammatory joint disease, including sequalae of viral infections
6. Suspected or documented allergy or hypersensitivity to cobalt, chromium, nickel or other metals
7. History of keloid, hypertrophic or contracture scaring
8. Propensity for restrictive scar formation or adhesions with prior procedures

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-03 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from device- and procedure-related Subsequent Surgical Interventions | 5 years post-implantation

SECONDARY OUTCOMES:
WOMAC Pain | 5 years
  Percent of subjects meeting clinically meaningful improvement (defined as ≥ 10-point change from baseline) Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used for evaluation of pain. The responses to each question are summed and the resultant scores are transformed to a 0-100 scale. A WOMAC score of zero (0) represents no knee problems and one hundred (100) represents extreme knee problems.
WOMAC Function | 5 years
  Percent of subjects meeting clinically meaningful improvement (defined as ≥ 10-point change from baseline).
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) was used for evaluation of function. The responses to each question are summed and the resultant scores are transformed to a 0-100 scale. A WOMAC score of zero (0) represents no knee problems and one hundred (100) represents extreme knee problems.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Crawford, MD, Principal Investigator — Oregon Health and Science University
Locations (3):
- United States (3):
  - Weiss Orthopedics, Sonoma, California
  - Oregon Health and Science University, Portland, Oregon
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No